CLINICAL TRIAL: NCT00012025
Title: Phase II Trial Of Fulvestrant (Faslodex) In Women With Metastatic Breast Cancer And Failure on Aromatase Inhibitor Therapy
Brief Title: ICI 182780 in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0032; CDR0000068473 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fulvestrant (Experimental): Patients receive fulvestrant intramuscularly on day 1. Courses repeat approximately every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months for 5 years or until disease progression. After disease progression, patients are followed every 3 months for 2 years and then every 6 months for 3 years.
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: fulvestrant

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using ICI 182780 may fight breast cancer by blocking the activity of estrogen in the tumor cells.

PURPOSE: Phase II trial to study the effectiveness of ICI 182780 in treating patients who have metastatic breast cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and partial objective response rate and duration of response in women with metastatic breast cancer who have failed aromatase inhibitor therapy treated with fulvestrant.
* Determine the time to disease progression and overall survival of women treated with this drug.
* Determine the toxicity of this drug in these women.

OUTLINE: Patients receive fulvestrant intramuscularly on day 1. Courses repeat approximately every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 5 years or until disease progression. After disease progression, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Progressive local-regional or metastatic disease
  * Unconfirmed new or progressive multiple pulmonary nodules or unequivocal radiographic evidence of multiple bone metastases allowed
* At least 1 measurable lesion

  * At least 20 mm by CT scan or MRI OR at least 10 mm by spiral CT scan
  * Nonmeasurable disease includes the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusions
    * Lymphangitis cutis/pulmonis
    * Inflammatory breast disease
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* Disease progression after prior third-generation aromatase inhibitor (e.g., anastrozole, exemestane, letrozole, or vorozole)

  * Failed no more than 1 prior additive hormonal therapy (e.g., aromatase inhibitor with or without tamoxifen)

    * Disease recurrence identified no more than 12 months since the last prior adjuvant tamoxifen treatment
    * Oophorectomy, ovarian radiotherapy, and luteinizing hormone-releasing hormone (LH-RH) analogs not considered hormonal therapy regimens
* No brain or leptomeningeal metastases
* No hepatic metastases involving more than one-third of the liver
* No symptomatic pulmonary lymphangitic disease
* Evidence of hormone sensitivity as defined by:

  * Relapse after at least 12 months of adjuvant hormonal treatment
  * Tumor remission or stabilization before progression for at least 6 months after prior hormonal therapy for advanced disease
* Postmenopausal as defined by one of the following:

  * At least 12 months since last menstrual period
  * 4-11 months since last menstrual period and follicle-stimulating hormone (FSH) in the postmenopausal range
  * Prior castration and castrate FSH levels within the postmenopausal range
  * Hysterectomy without oophorectomy (FSH in postmenopausal range if age 60 and under)
* Hormone receptor status:

  * Estrogen-receptor and/or progesterone-receptor positive

    * At least 10 fmol/mg cytosol protein OR
    * Positive by immunohistochemistry

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* See Disease Characteristics
* Postmenopausal

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* No history of bleeding diathesis

Hepatic:

* See Disease Characteristics
* Bilirubin no greater than 0.8 mg/dL above upper limit of normal (ULN)
* INR no greater than 1.6
* No hepatitis B or C
* No severe hepatic impairment

Renal:

* Calcium no greater than 10% above ULN
* Creatinine no greater than 1 mg/dL above ULN
* No severe renal impairment

Cardiovascular:

* No unstable or uncompensated cardiac condition

Pulmonary:

* No unstable or uncompensated respiratory condition

Other:

* HIV negative
* No AIDS
* No other severe condition or systemic disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior trastuzumab (Herceptin) allowed

Chemotherapy:

* Prior adjuvant chemotherapy allowed
* No more than 1 prior chemotherapy regimen for metastatic disease

Endocrine therapy:

* See Disease Characteristics
* More than 4 weeks since prior estrogen replacement therapy
* More than 3 months since prior LH-RH analogs
* No other prior additive hormonal therapy except third-generation aromatase inhibitors or tamoxifen

Radiotherapy:

* See Disease Characteristics
* Concurrent radiotherapy for control of bone pain or other reasons due to established bone lesions allowed if radiotherapy field is no more than 30% of bone marrow

Surgery:

* See Disease Characteristics

Other:

* More than 4 weeks since prior investigational drug for breast cancer
* No concurrent long-term warfarin
* Concurrent bisphosphonates allowed if dose stable
* Concurrent long-term antiplatelet therapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-05; Primary Completion 2006-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
objective response rate | Up to 10 years

SECONDARY OUTCOMES:
overall survival | Up to 10 years
time to disease progression | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: James N. Ingle, MD, Study Chair — Mayo Clinic
Locations (25):
- United States (24):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Carle Foundation Hospital - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Ingle JN, Suman VJ, Rowland KM, Mirchandani D, Bernath AM, Camoriano JK, Fishkin PA, Nikcevich DA, Perez EA; North Central Cancer Treatment Group Trial N0032. Fulvestrant in women with advanced breast cancer after progression on prior aromatase inhibitor therapy: North Central Cancer Treatment Group Trial N0032. J Clin Oncol. 2006 Mar 1;24(7):1052-6. doi: 10.1200/JCO.2005.04.1053. PMID 16505423
- [Result] Ingle JN, Rowland KM, Suman VJ, et al.: Evaluation of fulvestrant in women with advanced breast cancer and progression on prior aromatase inhibitor therapy: a phase II trial of the North Central Cancer Treatment Group. [Abstract] Breast Cancer Res Treat 88 (1): A-409, 2004.